CLINICAL TRIAL: NCT05855265
Title: Response Of RTOG Scale and Dermoscopy to Photon Therapy Face Mask on Dermatitis Post Head and Neck Radiotherapy
Brief Title: Photon Therapy Face Mask on Dermatitis Post Head and Neck Radiotherapy
Acronym: dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khadra Mohamed Ali (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Khadra Mohamed Ali, assisst professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 264200
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Cancers - Nasopharyngeal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (SG) (Experimental): The patients in study group treated with photon therapy (3x/week) for 6 weeks with a total of 18 sessions and Routine methods of nursing were given during radiotherapy including health education, skin self-care, and skin protective agent .The severity of skin reactions was assessed by the criteria of the Radiation Therapy Oncology Group (RTOG) and dermoscopy for both groups were recorded.
  Interventions: Device: photon therapy face mask
- control group (CG) (Experimental): Routine methods of nursing were given during radiotherapy including health education, skin self-care, and skin protective agent for control groups CG.The severity of skin reactions was assessed by the criteria of the Radiation Therapy Oncology Group (RTOG) and dermoscopy for both groups were recorded.
  Interventions: Device: photon therapy face mask

INTERVENTIONS:
Device: photon therapy face mask — In this study the patients were randomly assigned into two equal groups after agreeing to participate through signing an informed consent.,Out of 70 identified Nasopharyngeal tumor receiving radiotherapy, only 60 subjects completed the full requirements of the study,Participant's age ranged from 30-60 yearsThe subjects in control group (CG) were treated with their medical treatment in addition to routine methods of nursing were given during radiotherapy including health education, skin self-care, and skin protective agent. 0.9% normal saline cotton balls will be used to gently clean the wound and remove necrotic tissue, and the wound was dried with sterile gauze.
  The subjects in study group (SG) were received photon therapy during radiotherapy treatment. In addition to medical treatment and routine methods of nursing,

SUMMARY:
A randomized controlled trial (RCT), 60 HNC patients who underwent radiotherapy (RT) with or without chemotherapy represented the sample of the study. They were assigned randomly into two equal groups, control group (CG) and study group (SG). Routine methods of nursing were given during radiotherapy including health education, skin self-care, and skin protective agent for both groups CG and SG. The patients in study group treated with photon therapy (3x/week) for 6 weeks with a total of 18 sessions. The severity of skin reactions was assessed by the criteria of the Radiation Therapy Oncology Group (RTOG) and dermoscopy for both groups were recorded.

DETAILED DESCRIPTION:
This current study will be designed to prove the effect of photon therapy face mask on dermatitis post radiotherapy in patient with head and neck cancer. The measurements procedures will be conducted two times, before treatment application (pre-treatment) and after six weeks of treatment application (post-treatment). RTOG SCALE will be used to asset the patient before and after end of therapeutic procedures. Therapeutic intervention for the study was started at the same time for all groups of the study as following; Photon therapy will be applied from the first until the last day of RT (3×/week, 14 sessions). During the Photon therapy sessions, the whole irradiated area will be treated with 630 nm LED phototherapy. Treatment time will be 3 sessions per week for 30 min. set at 4 J/cm2 . Patients who will receive photon therapy during radiotherapy treatment within 2 weeks in addition to medical treatment and routine methods of nursing will be given during radiotherapy, including health education, skin self-care, and skin protective agent. 0.9% normal saline cotton balls will be used to gently clean the wound and remove necrotic tissue, and the wound will be dried with sterile gauze.

ELIGIBILITY:
Inclusion Criteria:

* All patients were free from any skin diseases, All patients enrolled to this study signed their informed consent,All the patients who had Nasopharyngeal tumor receiving radiotherapy who participated in this study, diagnosed by an oncologist and confirmed by MRI, C.T and laboratory investigations).

Exclusion Criteria:

* patients with communication disorders, patients who were unwilling to take part in this treatment, patients with tumor recurrence, patients with tumor stage 3 or more and patients with skin diseases

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Radiation Therapy Oncology Group/European Organization for Research and Treatment of Cancer (RTOG/EORTC) | once per week during treatment period for 6 weeks
  The assessment of dermatitis by RTOG scale was conducted by the physician once per week during treatment period . The grading of the RTOG scale : Grade 0: no change, Grade 1: Slight atrophy; pigmentation change; some hair loss, Grade 2: Patch atrophy; moderate telangiectasia; total hair loss, Grade 3: Marked atrophy; gross telangiectasia and Grade 4: ulcer, bleeding, and necrosis
Dermoscopic score | 3 months
  Erythema was graded from 0 to 3 (Figure 1), where 0 5= no erythema, 1 = faint erythema, 2 = moderate erythema, and 3 = erosion. Scaling was graded from 0 to 2, where 0 = no scaling, 1=moderate scaling, and 2 = severe scaling. Similarly, pigmentation was graded from 0 to 2, where 0 = no pigmentation, 1= moderate pigmentation, and 2 = severe pigmentation. The score was then calculated by the addition of the aforementioned grades (erythema + scaling + pigmentation) to produce a score ranging from 0 to 7, where 7 is the most severe and 0 represents no erythema, no scaling, and no pigmentation. For assessment of therapeutic response, the dermoscopic score of a fixed area, calculated 2 weeks after the first radiation therapy session, four weeks after the first radiation therapy session and after finishing radiation therapy sessions, was compared with the baseline dermoscopic score of the same area.

CONTACTS AND LOCATIONS:
Overall Officials: Ali, Principal Investigator — assist professor - department of physical therapy for surgery - Cairo university
Locations (1):
- faculty of physical therapy , Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The purpose of this study was to evaluate the effect of photon therapy in reducing the dermatitis during and post radiotherapy in patients with head and neck tumors. A randomized controlled trial (RCT), 60 HNC patients who underwent radiotherapy (RT) with or without chemotherapy represented the sample of the study. They were assigned randomly into two equal groups, control group (CG) and study group (SG). Routine methods of nursing were given during radiotherapy including health education, skin self-care, and skin protective agent for both groups CG and SG. The patients in study group treated with photon therapy (3x/week) for 6 weeks with a total of 18 sessions. The severity of skin reactions was assessed by the criteria of the Radiation Therapy Oncology Group (RTOG) and dermoscopy for both groups were recorded.
Supporting Information: Study Protocol, ICF
Time Frame: Photon therapy was applied from the beginning of the treatment till the end of the treatment with radiation therapy (three times per week, for six weeks with a total of 18 sessions). During the photon therapy sessions, the irradiated area was treated. Treatment wavelength parameter was 630 nm LED phototherapy 15. Treatment time per session was 20 min . data available at May 2022.
Access Criteria: inclusion Criteria:
  The subject selection was according to the following criteria:
  * Age ranged between 30-60 years.
  * Male and female patients participated in the study.
  * All the patients had nasopharyngeal type of head and neck cancers were receiving radiation therapy (IMRT).
  * All patients were free from any skin diseases.
  * All patients enrolled to this study signed their informed consent.
  Exclusion Criteria:
  The potential participants were excluded if they met one of the following criteria:
  * Patients with communication disorders.
  * Patients who were unwilling to take part in this treatment.
  * Patients with skin diseases.
  * patients with tumor recurrence.
  * patients with tumor stage 3 or more.